CLINICAL TRIAL: NCT03980587
Title: Exploratory Study of Molecular Characterization in Patients With Metastatic Germ Cell Tumours Refractory/Resistant to Platinum Treatment
Acronym: EMIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: University College London (UCL) Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4911
Record Dates: First submitted 2019-04-29; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-03

CONDITIONS: Testicular Germ Cell Tumor
Keywords: ctDNA
MeSH Terms: conditions — Testicular Germ Cell Tumor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood samples have been collected and stored in Royal Marsden Biobank. Archived tumour samples may also be used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To establish whether circulating tumour DNA is detectable in the plasma of patients with platinum refractory/resistant Germ Cell Tumours
2. If ctDNA is detectable, perform exploratory analyses to:

   1. Describe the molecular aberrations in plasma from metastatic GCTs with platinum refractory/resistant disease
   2. Describe aberrations detected in sequential detected in sequential samples form the same individual patient and evaluate whether there are hyposthesis-generating changes that temporarily associate with clinical resistance.

DETAILED DESCRIPTION:
This project will study the plasma of patients who have metastatic GCTs with platinum refractory/resistant disease in order to establish if ctDNA is detectable and then analyse the molecular aberrations. Archival diagnostic tissue will be recalled (this is the tissue used to make the initial diagnosis of testicular cancer). Excess tissue acquired from clinically mandated prospective biopsies will be stored and plasma which has been collected at a maximum of 15 time-points per year will be analysed. Clinical data will be accessed to make clinically meaningful associations with plasma and tissue molecular aberrations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed metastatic GCT refractory/resistant to platinum treatment
* Patients who have signed the 'Tissues for Research' consent form at the Royal Marsden Hospital and have blood samples stored in the RMH Biobank.
* Patients with no prior or current non-testicular invasive malignancy within the last 3 years, other than non-melanoma skin cancer or NCCN low risk prostate cancer (pT1 or pT2a Gleason ≤ 6, PSA ≤ 10 and ≤ 1cc total volume)

Exclusion Criteria:

* n/a

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will have consented to the collection and storage of blood samples and archival tissue at the RMH bio-bank. Testicular cancer management is focused in a single multidisciplinary clinic (Sutton Friday AM) and is the centre for follow up of these patients. We propose to initially analyseclinical material from 18 patients who have attended this clinic. To meet our primary objective, patient samples will be selected based on the burden of metastatic tumour in the patient at the time of the blood sample. Samples will be selected from patients at the latest available time-point in their disease process where the disease burden was at its highest.
  The minimum sample requirement for our primary and secondary objectives is a blood sample taken during at least one timepoint. However if there are an excess of patients with bloods samples collected when metastatic disease burden is at its highest, patient samples will be preferentially selected if they have sequential samples.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Circulating DNA in plasma is measurable | 1 year
  Measurement of plasma of patients with platinum refractory/resistant germ cell tumours
Exploratory analysis of circulating DNA | 1 year
  1. describe the molecular aberrations in plasma from metastatic germ cell tumours with platinum resistant/refractory disease
  2. Describe aberrations detected in sequential samples from the same indivivdual patient and evaluate whether there are hypothesis-generating changes that temporally associate with clinical resistance

CONTACTS AND LOCATIONS:
Overall Officials: Alison Reid, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided